CLINICAL TRIAL: NCT06258837
Title: Treatment of Obstructive Sleep Apnea With Personalized Surgery in Children With Small Tonsils
Acronym: TOPS-ST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Derek Lam, MD, MPH, Professor, Otolaryngology-Head and Neck Surgery, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00027270
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Otolaryngological Disease; Obstructive Sleep Apnea
MeSH Terms: conditions — Otorhinolaryngologic Diseases; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from pediatric otolaryngology clinics. The study will be introduced to caregivers of children with small tonsils and a history of sleep disordered breathing/OSA who are referred for surgery and meet the inclusion and exclusion criteria noted. If current or recent PSG testing demonstrates OSA, they will be invited to participate.
  Randomization will be done. Patients will be randomized to either the personalized DISE-directed surgery or the standard AT after collection of baseline measures and pre-op PSG. Allocation will be made by using a computer-generated randomization scheme. Caregivers will be advised of the outcomes and risks of different surgical procedures included in DISE-directed surgery and informed consent will be obtained. All patients will be planned for overnight observation to monitor for safety and perioperative complications.
Who Masked: Outcomes Assessor
Masking Description: It is not practical or feasible to maintain blinding among the surgeons performing the procedures or the clinical staff caring for patients in the perioperative setting. Given this, it is unlikely that blinding could be maintained among parents or caregivers of patients, therefore there will be no attempt to blind caregivers to the treatment assignment. However, the sleep medicine collaborators who will be reviewing and scoring postoperative PSGs will be instructed not to review the medical record so as to ensure blinding to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug-Induced Sleep Endoscopy (Experimental): DISE will be performed at the time of surgery under the same sedation. The decision on specific surgical approach will be made at that time based on DISE findings. Prior to intubation, patients will be sedated with either a propofol infusion or a combination of ketamine and dexmedetomidine. Once adequate sedation is achieved, endoscopy will be performed using a flexible endoscope advanced through the nose. The nasal airway will be evaluated on both sides, then the endoscope will be advanced into the pharynx. The degree of obstruction is scored on a 3-point rating scale. Participants randomized to DISE-directed surgery will undergo one or more potential procedures in a single surgery. Caregivers will be consented for all possible procedures with the understanding that only those needed based on DISE will be performed. Importantly, these procedures are all established treatments with published outcomes data.
  Interventions: Procedure: DISE-Directed Surgery
- Adenotonsillectomy (Active Comparator): Adenotonsillar hypertrophy is the most common risk factor for OSA in children, and adenotonsillectomy (AT) is the first line treatment. An adenotonsillectomy is an operation to remove both the adenoids and tonsils.
  Interventions: Procedure: Adenotonsillectomy

INTERVENTIONS:
Procedure: DISE-Directed Surgery — Participants randomized to DISE-directed surgery will undergo one or more potential procedures in a single surgery (i.e. DISE and subsequent sleep surgery performed) concurrently under the same general anesthetic), depending on anatomic assessment.
  Other Names: sleep endoscopy
  Arms: Drug-Induced Sleep Endoscopy
Procedure: Adenotonsillectomy — Tonsil and/or adenoid removal
  Other Names: AT
  Arms: Adenotonsillectomy

SUMMARY:
The purpose of this study is to compare the effectiveness of a novel personalized surgical approach to the standard AT in children with small tonsils (ST). This will be accomplished by randomizing children with ST and OSA to one of these two treatments and comparing outcomes after 6 months. It is the investigators' central hypothesis that a personalized drug-induced sleep endoscopy (DISE)-directed surgical approach that uses existing procedures to address the specific fixed and dynamic anatomic features causing obstruction (ie, anatomic endotypes) in each child with ST will perform better than the currently recommended standard first line approach of AT. This novel approach may improve OSA outcomes and reduce the burden of unnecessary AT or secondary surgery for persistent OSA after an ineffective AT. To test this hypothesis, the investigators propose to study children aged 2-17 years with small tonsils and OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is common in children with an estimated prevalence of 1-6%. Untreated pediatric OSA is associated with hypertension, autonomic dysfunction, attention-deficit / hyperactivity disorder, neurocognitive deficits, poor school performance, poor quality of life, and a >200% increase in health care utilization compared to controls. Adenotonsillar hypertrophy is the primary risk factor for pediatric OSA, and adenotonsillectomy (AT) is the recommended first line treatment. However, the prevalence of persistent OSA after AT has been reported to be at least 20% among children with large tonsils, indicating that AT may not be the optimal intervention in all cases. Although the prevalence of small tonsils in children with OSA symptoms is up to 70%, there is currently no clear evidence on the outcome of AT in children with small tonsils. It has been shown that clinic assessments of tonsil size do not correlate with OSA severity or response to AT, leaving confusion about how best to treat OSA in children with small tonsils. This knowledge gap represents an opportunity to apply a personalized treatment approach and improve outcomes.

DISE entails passage of a flexible endoscope through the nose into the pharynx and enables direct observation of the sites and patterns of upper airway obstruction during sedated sleep. DISE was developed to guide surgical decisions in adult OSA, and in recent years has also been used to design personalized surgical interventions in children. To help standardize DISE assessments, the investigators previously developed and validated the DISE Rating Scale in children based on ordinal ratings of maximal airway obstruction (none, partial, complete) at six anatomic sites from the nose to the larynx.

The investigators also demonstrated that DISE ratings of adenotonsillar obstruction during sedated sleep are strongly associated with both OSA severity and response to AT, unlike clinic assessments of tonsil size. The investigators' preliminary data and other published studies have identified a high prevalence of non-adenotonsillar obstruction that can occur at the nose, palate, base of tongue, and larynx. Surgery that is tailored to the specific anatomic sites of obstruction observed during DISE may improve pediatric OSA outcomes, but existing studies are small, uncontrolled case series in heterogeneous study populations. There are no trials directly comparing AT and DISE-directed surgery in the common scenario of surgically naïve children with small tonsils.

The purpose of this study is to compare the effectiveness of a novel personalized surgical approach to the standard AT in children with small tonsils (ST). This will be accomplished by randomizing children with ST and OSA to one of these two treatments and comparing outcomes after 6 months. It is the investigators' central hypothesis that a personalized drug-induced sleep endoscopy (DISE)-directed surgical approach that uses existing procedures to address the specific fixed and dynamic anatomic features causing obstruction (i.e., anatomic endotypes) in each child with ST will perform better than the currently recommended standard first line approach of AT. This novel approach may improve OSA outcomes and reduce the burden of unnecessary AT or secondary surgery for persistent OSA after an ineffective AT. To test this hypothesis, the investigators propose to study children aged 2-17 years with small tonsils and OSA.

ELIGIBILITY:
To be in the study:

* Child has a diagnosis of moderate to severe OSA diagnosed by PSG (oAHI ≥ 5).
* Child age is 2.00 to 17.99 years of age.
* Child has small tonsils (Brodsky 1+ or 2+) noted during routine physical exam.
* Caregiver can provide signed and dated consent and is 18 years of age or older at the time of consent.
* Caregiver can speak, read, and write in English or Spanish.
* Caregiver is primary caretaker of the child.
* Child is not expecting their own child.
* Child is eligible for surgical treatment

Cannot be in the study if:

* Child has history of previous tonsillectomy, tonsillotomy, or partial tonsillectomy.
* Child has any contraindication to surgery (e.g. bleeding disorders).
* Child has significant cardiopulmonary comorbidity besides OSA requiring supplemental oxygen, subglottic or tracheal stenosis, tracheostomy dependence.
* Child has a genetic abnormality, Down syndrome, neuromuscular disorder, craniofacial anomaly.
* Caregiver is unwilling or unable to comply with study procedures.
* Child is or plans to become a parent themselves.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Polysomnography Measures: Obstructive Apnea-Hypopnea Index (oAHI) at 6 months | 6 month follow up sleep study (after surgery)
  Objective results from sleep studies (polysomnography): Obstructive Apnea-Hypopnea Index (oAHI): 6 months follow up sleep study difference from baseline sleep study. Higher scores indicate higher disease burden. Scores can range from zero to two hundred.
Change from Baseline Polysomnography Measures: Total Apnea-Hypopnea Index (AHI) at 6 months | 6 month follow up sleep study (after surgery)
  Objective results from sleep studies (polysomnography): Total Apnea-Hypopnea Index: 6 months follow up sleep study difference from baseline sleep study. Higher scores indicate higher disease burden. Scores can range from zero to two hundred.
Change from Baseline Polysomnography Measures: REM Apnea-Hypopnea Index (REM AHI) at 6 months | 6 month follow up sleep study (after surgery)
  Objective results from sleep studies (polysomnography): REM Apnea-Hypopnea Index REM AHI: 6 months follow up sleep study difference from baseline sleep study. Higher scores indicate higher disease burden. Scores can range from zero to two hundred.
Change from Baseline Polysomnography Measures: minimum Oxygen saturation (SpO2) at 6 months | 6 month follow up sleep study (after surgery)
  Objective results from sleep studies (polysomnography): Minimum Oxygen Saturation (Min SpO2): 6 months follow up sleep study difference from baseline sleep study. Lower scores indicate higher disease burden. Scores range from 0-100, although neither extreme is actually seen in patients.
Change from Baseline Polysomnography Measures: Oxyhemoglobin desaturation ≥ 3% Index (desat index) at 6 months | 6 month follow up sleep study (after surgery)
  Oxyhemoglobin desaturation ≥ 3% Index: 6 months follow up sleep study difference from baseline sleep study. Higher scores mean higher disease burden. Mild desaturation (< 5.0 events/h), moderate desaturation (≥ 5.0 events/h and < 10.0 events/h), and severe desaturation (≥ 10.0 events/h).
Change from Baseline Polysomnography Measures: Percent Total Sleep Time with ETCO2 > 50 mmHg at 6 months | 6 month follow up sleep study (after surgery)
  % Total Sleep Time with ETCO2 > 50 mmHg: 6 months follow up sleep study difference from baseline sleep study. Higher scores mean higher disease burden. Scores range from 0-100.
Change from Baseline Polysomnography Measures: Max End Tidal CO2 (ETCO2) at 6 months | 6 month follow up sleep study (after surgery)
  Max End Tidal CO2 (ETCO2): 6 months follow up sleep study difference from baseline sleep study. Higher scores mean higher disease burden. Normal is 35-40 mmHg.

SECONDARY OUTCOMES:
Change in Obstructive Sleep Apnea (OSA)-18 Questionnaire score | 6 month follow up
  Disease specific quality of life measure: 18 questions, scores range from 18-126; higher scores means higher disease burden
Change in Generic PedsQL (Pediatric Quality of Life) Questionnaire score | 6 month follow up
  Generic quality of life measure: an age specific questionnaire with 23 questions (scores range from 0-100); higher scores indicate better quality of life.
Change in Generic PedsQL (Pediatric Quality of Life) Questionnaire answers | 6 month follow up
  Quality of life: questionnaire results by individual question. Adjusted scores range from 0-100; higher scores indicate better quality of life.
Total Drug induced sleep endoscopy (DISE) score | At time of surgery
  Subjective ratings of degree of obstruction at 6 levels of the upper airway, done by surgeon. Scores range from 0 to 12. Higher scores means more breathing obstruction, or more disease burden.
Adverse Events | 24 hour period after surgery
  Did any adverse events occur in the post-operative time frame? This is a yes/no question, looking at the following outcomes: dehydration and poor oral intake due to post-operative pain, post-tonsillectomy hemorrhage, and respiratory compromise.
Change in Child Behavior Checklist (CBCL) Questionnaire answers | Baseline versus 6 month follow up
  Assesses behavioral and emotional problems: questionnaire results by total score and by "syndrome scale scores". Adjusted norms scores range from 0.0-1.0; higher scores indicate greater problems.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Lam, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to researchers who are not primary researchers on this study.